CLINICAL TRIAL: NCT06903871
Title: A Prospective, Randomized, Open-label, Controlled Clinical Study Comparing Toripalimab Adjuvant Therapy Versus Clinical Observation in Subjects With Resected Esophageal Squamous Cell Carcinoma Who Achieved Pathological Complete Response (pCR)
Brief Title: Toripalimab Adjuvant Therapy in Subjects With Resected Esophageal Squamous Cell Carcinoma Who Achieved Pathological Complete Response (pCR)
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Hebei Medical University Fourth Hospital (Other)
Responsible Party: Principal Investigator, JunFeng Liu, MD, Director of thoracic surgery, Hebei Medical University Fourth Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HebeiJLiu-ESCC-2025
Record Dates: First submitted 2025-03-21; First posted 2025-04-01 (Actual); Last update posted 2025-04-01 (Actual); Status verified 2025-03

CONDITIONS: Esophageal Squamous Cell Carcinoma Stage II; Esophageal Squamous Cell Carcinoma Stage III
MeSH Terms: conditions — Esophageal Squamous Cell Carcinoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Toripalimab (Experimental)
  Interventions: Drug: TORIPALIMAB INJECTION(JS001 )
- control (No Intervention)

INTERVENTIONS:
Drug: TORIPALIMAB INJECTION(JS001 ) — Participants will receive toripalimab 240 mg IV once every 3 weeks. Treatment continued until disease progression, death, unacceptable toxicity, investigator decision, withdrawal, or completion of 1 years of treatment, whichever occurred first.
  Arms: Toripalimab

SUMMARY:
The goal of this clinical trial is to assess the 1-year DFS rate of toripalimab adjuvant therapy in participants with resected esophageal squamous cell carcinoma (ESCC) who achieved pCR. The main questions it aims to answer are:

* The toripalimab adjuvant therapy could impove the 1-year DFS rate in participants with rescted ESCC who achieved pCR?
* Is this treatment regimen safe? Researchers will compare toripalimab adjuvant therapy to clinical observation to see if toripalimab could improve the 1-year DFS rate.

Participants will receive toripalimab 240 mg IV once every 3 weeks for one year or clinical observation.

ELIGIBILITY:
Inclusion Criteria:

* Stage II or III esophageal cancer with histologically confirmed predominant squamous cell carcinoma at initial diagnosis;
* Subjects must complete preoperative neoadjuvant therapy (unlimited treatment regimen) before being assigned to treatment and then undergo surgery;
* Subjects must undergo complete resection (R0), be surgically determined to be disease-free and have a negative margin on the resected specimen, defined as no viable tumor within 1 mm of the proximal, distal, or surrounding resection boundary;
* Subjects must have no residual pathology, the primary tumor is pCR, and the pathology report of the resected lymph nodes is ypN0;
* ECOG performance status of 0 or 1;
* The laboratory test meet the following requirements:

Bone marrow function: neutrophils ≥ 1.5×10(9)/L, platelets ≥ 100×10(9)/L, hemoglobin ≥ 90 g/L Liver function：Total bilirubin ≤ 1.5 x ULN；AST and ALT ≤ 3 x ULN Renal function：Cr ≤ 1.5 x ULN，Ccr ≥ 50 ml/min.

Exclusion Criteria:

* Subjects with stage M1 resectable disease；
* Received treatments for resected esophageal cancer (e.g., immunotherapy , chemotherapy, targeted therapy, radiotherapy, or biologic therapy);
* Known to be allergic, highly sensitive or intolerable to research-related drugs or excipient
* In the past 5 years, there were other malignant tumors, melanoma skin cancer or ervical carcinoma in situ were excepted.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 190 (Estimated)
Dates: Start 2025-04-01 (Estimated); Primary Completion 2029-03-01 (Estimated); Study Completion 2030-03-01 (Estimated)

PRIMARY OUTCOMES:
1-year Disease free survival rate | 1 year

SECONDARY OUTCOMES:
1, 2, 3 years overall survival rates | 3 years
Distant metastasis-free survival | 2 years
Number of Participants with Adverse Events as a Measure of Safety and Tolerability | 1.5 years
  The incidences of adverse events were calculated according to the National Cancer Institute Cancer Common Toxicity Criteria, version 5.0.

CONTACTS AND LOCATIONS:
Locations (1):
- Hebei Medical University Fourth Hospital, Shijiazhuang, Hebei, China